CLINICAL TRIAL: NCT03151629
Title: International Registry for Men With Advanced Prostate Cancer (IRONMAN)
Acronym: IRONMAN
Status: Recruiting | Type: Observational
Sponsor: Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: c16-170
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Castrate Resistant Prostate Cancer
  Interventions: Other: Standard of Care
- Hormone Sensitive Prostate Cancer
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Drugs routinely administered for metastatic prostate cancer per local standard.

SUMMARY:
Our intent is to establish the International Registry to Improve Outcomes in Men with Advanced Prostate Cancer (IRONMAN) as a prospective, international cohort of minimum 5,000 men with advanced cancer, including men with mHSPC and M0/M1 CRPC. The goal is to establish a population-based registry and recruit patients across academic and community practices from Australia, Barbados, Brazil, Canada, Ireland, Jamaica, Kenya, Nigeria, Norway, Spain, South Africa, Sweden, Switzerland, the United Kingdom (UK), and the United States (US). Target accrual number and number of participating sites are subject to change based on accrual, funding, and interest in participation by other international sites. This cohort study will facilitate a better understanding of the variation in care and treatment of advanced prostate cancer across countries and across academia and community based practices.

Detailed data will be collected from patients at study enrollment and then during follow-up, for a minimum of five years. Patients will be followed prospectively for overall survival, clinically significant adverse events, comorbidities, changes in cancer treatments, and PROMs.

PROMs questionnaires will be collected at enrollment and every three months thereafter.

Physician Questionnaires will be collected from all participating sites at patient enrollment, time of first change in treatment and/or one year follow-up, at each subsequent change of treatment, and discontinuation of treatment.

As such, this registry will help identify the treatment sequences or combinations that optimize overall survival and PROMs for men with mHSPC and M0/M1 CRPC. By collecting blood at enrollment, time of first change in treatment and/or one year follow-up (plasma, cell free DNA, buffy coat / RNA), this registry will further identify and validate molecular phenotypes of disease that predict response and resistance to specific therapeutics. Additionally, every effort will be made to collect blood specimen at each subsequent change in treatment due to progression of disease. When feasible, existing tumor tissue may be collected for correlation with described blood based studies. All samples will be used for future research. This cohort study will provide the research community with a unique biorepository to identify biomarkers of treatment response and resistance.

ELIGIBILITY:
• Willing and able to provide written informed consent and privacy authorization for the release of personal health information.

NOTE: Privacy authorization may be either included in the informed consent or obtained separately.

* Males 21 years of age and above
* Histological or cytological confirmed prostate adenocarcinoma from TRUS biopsy, radical prostatectomy or TURP Or Documented histopathology or cytopathology of prostate adenocarcinoma from a biopsy of a metastatic site Or Metastatic disease typical of prostate cancer (i.e., involving bone or pelvic lymph nodes or para-aortic lymph nodes) AND a serum concentration of PSA >20ng/mL at the time of initial prostate cancer diagnosis
* No previous diagnosis of a second, non-prostate malignancy that requires additional systemic therapy except cancer in situ of bladder and basal cell cancer of skin

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Study Population: Metastatic hormone sensitive prostate cancer (mHSPC): Prostate cancer patients diagnosed with histologically confirmed cancer with radiological evidence of metastatic disease and on ADT for no more than 90 days.
  Castration resistant prostate cancer (CRPC): Prostate cancer patients (with or without radiological evidence of metastatic disease) with a confirmed rising PSA (at least two measures) while on ADT or orchiectomy or castrate level of testosterone as determined by investigator.
  Prostate cancer patients with mixed histological types may participate in this Registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Practice Patterns | 5 years
  To describe the practice patterns of therapeutic agents for treatment of advanced prostate cancer internationally

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke Cancer Institute; Lorelei Mucci, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Phillip Kantoff, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (121):
- United States (48):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - University of Alabama- Tuscaloosa, Tuscaloosa, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Kishwaukee Cancer Center, DeKalb, Illinois
  - Delnor Cancer Center, Geneva, Illinois
  - Warrenville Cancer Center, Warrenville, Illinois
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Chesapeake Urology Associates, Towson, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - VA Western New York Healthcare System, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke Cancer Network, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Doylestown Health, Doylestown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Temple Health, Philadelphia, Pennsylvania
  - Reading Health System, West Reading, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - William Jennings Bryan Dorn VAMC, Columbia, South Carolina
  - Memphis VA Medical Center, Memphis, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (11):
  - Royal Brisbane & Women's Hospital, Herston, Brisbane
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Redland Hospital, Cleveland, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth Healthcare, Mount Waverley, Victoria
  - Australian Urology Associates, Melbourne
  - Australian Prostate Centre, Melbourne N.
- The University of the West Indies - Cave Hill Campus, Bridgetown, Barbados
- Brazil (6):
  - Tacchini Hospital, Bento Gonçalves, Rio Grande do Sul
  - Hospital Beneficência Portuguesa, Bela Vista, São Paulo
  - Instituto do Câncer e Transplante, Curitiba
  - Centro de Pesquisa em Oncologia, Porto Alegre
  - Centro Paulista de Oncologia, São Paulo
  - Instituto Câncer do Estado de São Paulo, São Paulo
- Canada (7):
  - Cross Cancer Institute (Alberta Health Services), Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
- Ireland (4):
  - Beacon Hospital, Dublin, Leinster
  - Tallaght University Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Sligo University Hospital, Sligo
- The University of the West Indies - Mona Campus, Kingston, Jamaica
- University of Nairobi, Nairobi, Kenya
- Nigeria (4):
  - Federal Medical Centre Abeokuta, Abeokuta
  - University of Ilorin Teaching Hospital, Ilorin
  - Lagos State University Teaching Hospital, Lagos
  - University of Maiduguri Teaching Hospital, Maiduguri
- Oslo University Hospital, Oslo, Norway
- South Africa (3):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Groote Schuur Hospital, Cape Town
- Spain (12):
  - Vall d'Hebron Institute of Oncology, Barcelona, Catalonia
  - Institut Catalá d'Oncologia Badalona, Badalona
  - Fundació Institut Mar d'Investigacions Mèdiques (Hospital del Mar)., Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet (Zaragoza), Zaragoza
- Sweden (3):
  - Skane University Hospital, Malmo, Skåne County
  - Orebro University Hospital, Örebro
  - Umea University Hospital, Umeå
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - Ente Ospedaliero Cantonale, Bellinzona
  - Kantonsspital Graubünden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen
  - Onkozentrum Zürich, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (13):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Lister Hospital, Stevenage, Hertfordshire
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Velindre Cancer Centre, Cardiff
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - Guys St Thomas NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - South Tyneside District Hospital, South Shields
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rencsok EM, Slopen N, McManus HD, Autio KA, Morgans AK, McSwain L, Barata P, Cheng HH, Dreicer R, Gerke T, Green R, Heath EI, Howard LE, McKay RR, Nowak J, Pileggi S, Pomerantz MM, Rathkopf DE, Tagawa ST, Whang YE, Ragin C, Odedina FT, Kantoff PW, Vinson J, Villanti P, Haneuse S, Mucci LA, George DJ; IRONMAN Registry. Pain and Its Association with Survival for Black and White Individuals with Advanced Prostate Cancer in the United States. Cancer Res Commun. 2024 Jan 8;4(1):55-64. doi: 10.1158/2767-9764.CRC-23-0446. PMID 38108490
- [Derived] Rencsok EM, Stopsack KH, Slopen N, Odedina FT, Ragin C, Nowak J, McSwain L, Manarite J, Heath E, George DJ, Kantoff PW, Vinson J, Villanti P, Haneuse S, Mucci LA; IRONMAN Registry. Experience with the US health care system for Black and White patients with advanced prostate cancer. Cancer. 2023 Aug 15;129(16):2532-2541. doi: 10.1002/cncr.34885. Epub 2023 May 28. PMID 37246339
- [Derived] McKay RR, Gold T, Zarif JC, Chowdhury-Paulino IM, Friedant A, Gerke T, Grant M, Hawthorne K, Heath E, Huang FW, Jackson MD, Mahal B, Ogbeide O, Paich K, Ragin C, Rencsok EM, Simmons S, Yates C, Vinson J, Kantoff PW, George DJ, Mucci LA. Tackling Diversity in Prostate Cancer Clinical Trials: A Report From the Diversity Working Group of the IRONMAN Registry. JCO Glob Oncol. 2021 Apr;7:495-505. doi: 10.1200/GO.20.00571. PMID 33835826